CLINICAL TRIAL: NCT00455845
Title: A Double Blind Randomized Controlled Trial to Study the Effectiveness of a Levonorgestrel Releasing Intrauterine Device for the Treatment of Pelvic Pain or Dysmenorrhea in the Patients Undergone Conservative Surgery for Pelvic Endometriosis
Brief Title: The Effectiveness of Lng IUD for Treatment of the Patient Undergone Conservative Surgery for Pelvic Endometriosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Associate Prof. Prasong Tanmahasamut, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 15/2007
Record Dates: First submitted 2007-04-03; First posted 2007-04-04 (Estimated); Last update posted 2011-03-02 (Estimated); Status verified 2007-04

CONDITIONS: Endometriosis; Pelvic Pain; Dysmenorrhea
Keywords: Endometriosis; Lng IUD
MeSH Terms: conditions — Endometriosis; Pelvic Pain; Dysmenorrhea

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 levonorgestrel IUD (Active Comparator)
  Interventions: Device: Levonorgestrel IUD
- 2 control (No Intervention)
  Interventions: Device: Levonorgestrel IUD

INTERVENTIONS:
Device: Levonorgestrel IUD — levonorgestrel IUD
  Other Names: Minera IUD

SUMMARY:
this study is to determine whether the frequency and severity of pelvic pain or dysmenorrhea are reduced in women with symptomatic endometriosis in whom a Lng IUD is inserted after operative laparoscopy compare with those treated with laparoscopic surgery only

DETAILED DESCRIPTION:
Endometriosis is a common cause of chronic pelvic pain.Laparoscopic surgery is often the treatment of choice for symptomatic disease and results are usually satisfactory but symptoms recur in 10-20% of treated women per year. Postoperative medical therapy has been controversial. Whereas some studies have observed a long pain free interval or higher pregnancy rates when surgical treatment is followed by an interval of medical suppressive treatment, numerous others have found no differences between the prevalence of recurrent pain or pregnancy rates 1-3 years after surgery treatment in women who did and did not receive postoperative medical treatment.Endometriosis is generally a localized disease but is currently managed with systemic medical therapies. The use of drugs administered locally and specifically aimed at pelvic organs could limit the metabolic impact without reducing antalgic efficacy.An intrauterine device releasing levonorgestrel, a potent 19-nortestosterone derivative progestin, can induce amenorrhea with a different modality with respect to standard regimens. The levonorgestrel intrauterine device (Lng-IUD) provides an alternative means of administering progestins.Some researchers reported the effectiveness of the Lng IUD in the patients with endometriosis.The primary objective of this study is to determine whether the frequency and severity of dysmenorrhea are reduced in women with symptomatic endometriosis in whom a Lng IUD is inserted after operative laparoscopy compare with those treated with laparoscopic surgery only.

The secondary objective is to compare about pain, bleeding, satisfaction and quality of life score between both groups

ELIGIBILITY:
Inclusion Criteria:

* women diagnosed endometriosis stage I-IV according to the revised American Society of Reproductive Medicine classification
* Moderate or severe pelvic pain or dysmenorrhea
* Undergoing conservative laparoscopic surgery

Exclusion Criteria:

* Patients who have uterine or adnexal anomalies other than endometriosis (chronic pelvic inflammatory disease, leiomyomas, endometrial polyps, genital malformations, pelvic varices)
* using treatments for endometriosis other than paracetamol,nonsteroid anti-inflammatory drugs or narcotic derivative in the 3 months before study entry
* Unable to perform conservative surgery
* Patients who have contraindications to Lng IUD as defined by the World Health Organization (2004).
* Patients who are unwilling to tolerate menstrual changes.
* Plan to have children within 1 year
* Unable to evaluate pain with visual analogue scale
* unwilling to participate this project

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2007-04; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
the frequency and severity of pelvic pain or dysmenorrhea | 12 months

SECONDARY OUTCOMES:
compare about pain, bleeding, satisfaction and quality of life score between both groups | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Prasong Tanmahasamut, M.D., Principal Investigator — Mahidol University
Locations (1):
- Mahidol University, Bangkoknoi, Bangkok, Thailand

REFERENCES:
- [Derived] Tanmahasamut P, Rattanachaiyanont M, Angsuwathana S, Techatraisak K, Indhavivadhana S, Leerasiri P. Postoperative levonorgestrel-releasing intrauterine system for pelvic endometriosis-related pain: a randomized controlled trial. Obstet Gynecol. 2012 Mar;119(3):519-26. doi: 10.1097/AOG.0b013e31824264c3. PMID 22314873